CLINICAL TRIAL: NCT03767335
Title: Open-label, Multicentre, Phase Ib Dose-escalation Study of MEN1611, a PI3K Inhibitor Combined With Trastuzumab With or Without Fulvestrant, in Subjects With PIK3CA Mutated HER2 Positive Locally Recurrent Unresectable (Advanced) or Metastatic (a/m) Breast Cancer Progressed to Anti-HER2 Based Therapy
Brief Title: MEN1611 With Trastuzumab (+/- Fulvestrant) in Metastatic Breast Cancer
Acronym: B-PRECISE-01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Menarini Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MEN1611-01; 2017-004631-36 (EudraCT Number)
Record Dates: First submitted 2018-12-05; First posted 2018-12-06 (Actual); Results first posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-04

CONDITIONS: Advanced or Metastatic Breast Cancer
Keywords: Advanced Breast Cancer; Metastatic Breast Cancer; PI3K inhibitor; HER2-positive
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Fulvestrant

STUDY DESIGN:
Intervention Model Description: Step 1 Dose escalation / Step 2 Cohort expansion in two selected breast cancer sub-populations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- MEN1611 (Experimental): MEN1611 + Trastuzumab +/- Fulvestrant
  Interventions: Drug: MEN1611; Drug: Trastuzumab; Drug: Fulvestrant

INTERVENTIONS:
Drug: MEN1611 — MEN1611 oral dose administered twice daily for a continuous 28-day cycle
Drug: Trastuzumab — Trastuzumab solution for infusion administered weekly via IV
Drug: Fulvestrant — Fulvestrant solution for injection administered monthly via IM (only for HR-positive postmenopausal women)

SUMMARY:
The main purpose of this open-label, dose-escalation, phase Ib study is to identify the appropriate dose of MEN1611 to be used in combination with Trastuzumab with/without Fulvestrant for the treatment of advanced or metastatic HER2-positive breast cancer

DETAILED DESCRIPTION:
This Phase Ib study will investigate the safety and anti-tumor activity of daily oral doses MEN1611 in combination with Trastuzumab with/without Fulvestrant in female and male patients affected by advanced or metastatic HER2-positive breast cancer. Fulvestrant will be added to the post-menopausal patients with hormone-sensitive disease.

MEN1611 is an investigational drug which blocks a protein called PI3K (phosphoinositide 3-kinase) involved in cancer cells growth. The Maximum Tolerated Dose (MTD) of MEN1611 given as single agent was assessed in a phase I trial in patients with advanced solid tumors.

This Phase IB will start with a dose escalation part (Step 1) to identify the MTD of MEN1611 given in combination with Trastuzumab with/without Fulvestrant.

The study will continue with a cohort expansion (Step 2) to investigate the anti-tumor activity of the selected MEN1611 dose level considered to be tolerable by a Safety Review Committee.

ELIGIBILITY:
Main Inclusion Criteria:

* Histologically confirmed invasive adenocarcinoma of the breast
* Known HER2+ breast cancer
* Advanced or metastatic breast cancer harbouring PIK3CA mutation on tissue sample
* > 2 lines of anti-HER2 based regimens with at least 1 regimen with trastuzumab
* Radiological documented evidence of progressive disease
* Life expectancy ≥ 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2

Main Exclusion Criteria:

* Previous treatment with PI3K inhibitors
* Brain metastases untreated, unless treated > 4 weeks and only if clinically stable and not receiving corticosteroids
* History of clinically significant bowel disease
* ≥ grade 2 diarrhoea
* History of significant, uncontrolled, or active cardiovascular disease
* Any serious and/or unstable pre-existing psychiatric or neurologic illness or other conditions that could interfere with patient's safety
* Not controlled diabetes mellitus (glycated haemoglobin [HbA1c] >7%) and fasting plasma glucose >126 mg/dL
* Concurrent chronic treatment with steroids, as immunosuppressant, or another immunosuppressive agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martine Piccart, MD PhD, Study Chair — Institute Jules Bordet - Boulevard De Waterloo 125 - B-1000 Brussels, Belgium
Locations (27):
- United States (3):
  - Holy Cross Hospital Inc., Fort Lauderdale, Florida
  - Detroit Clinical Research Center, Farmington Hills, Michigan
  - Washington University, St Louis, Missouri
- Belgium (3):
  - Cliniques Universitaires Saint-Luc, Brussels
  - Institut Jules Bordet, Brussels
  - UZ Leuven, Leuven
- France (6):
  - Centre Georges François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Institut Régional du Cancer de Montpellier, Montferrier-sur-Lez
  - ICO - Site René Gauducheau, Saint-Herblain
  - Institut Claudius Regaud Oncopole, Toulouse
  - Institut Gustave Roussy, Villejuif
- Italy (4):
  - Azienda Ospedaliero Universitaria Mater Domini, Catanzaro
  - Istituto Clinico Humanitas, Milan
  - Istituto Europeo di Oncologia (IEO), Milan
  - Ospedale San Raffaele, Milan
- Spain (7):
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Centro Integral Oncologico Clara Campal, Madrid
  - Hospital General Universitario Gregorio Marañon, Madrid
  - START Madrid Fundacion Jimenez Diaz, Madrid
  - Hospital Clínico Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen del Rocío, Seville
- United Kingdom (4):
  - Velindre Cancer Centre, Cardiff
  - Sarah Cannon Research Institute UK, London
  - University College London Hospitals, London
  - The Christie, Manchester

REFERENCES:
- [Derived] Fiascarelli A, Merlino G, Capano S, Talucci S, Bisignano D, Bressan A, Bellarosa D, Carrisi C, Paoli A, Bigioni M, Tunici P, Irrissuto C, Salerno M, Arribas J, de Stanchina E, Scaltriti M, Binaschi M. Antitumor activity of the PI3K delta-sparing inhibitor MEN1611 in PIK3CA mutated, trastuzumab-resistant HER2 + breast cancer. Breast Cancer Res Treat. 2023 May;199(1):13-23. doi: 10.1007/s10549-023-06895-2. Epub 2023 Mar 13. PMID 36913051

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 73 participants were screened for study eligibility, of which 11 were considered as screen failures.
Pre-assignment Details: The study included a Dose Escalation part and a Dose Expansion part. The Dose Escalation part of the study included Cohorts 1 and 2.
  It was prespecified that 3 participants who enrolled in Dose Expansion Cohort were to be included in the Dose-Limiting Toxicity (DLT) population. As prespecified, data were collected for the DLT population for the Maximum Tolerated Dose (MTD), DLT, Recommended Phase 2 Dose (RP2D) Outcome Measures,
Groups:
- Dose Escalation Cohort 1: Participants received low dose of MEN1611 twice daily administered in combination with trastuzumab once every 3 weeks ± fulvestrant once every 4 weeks.
- Dose Escalation Cohort 2: Participants received medium dose of MEN1611 twice daily administered in combination with trastuzumab once every 3 weeks ± fulvestrant once every 4 weeks.
- Dose Expansion Cohort: Participants received high dose of MEN1611 (Recommended Phase 2 dose [RP2D]) twice daily administered in combination with trastuzumab once every 3 weeks ± fulvestrant once every 4 weeks.
Period: Overall Study
Arm/Group | Dose Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Expansion Cohort
Started | 3 | 3 | 56
Received At Least 1 Dose of Study Drug | 3 | 3 | 56
DLT Population (DLT population consisted of all participants who received at least 80% of MEN1611 and 100% of trastuzumab and/or fulvestrant during 28 days after the first MEN1611 drug administration with a Safety Follow-up of 28 days after the first administration of the study treatment.) | 3 | 3 | 3
Completed (Only deaths notified as leading to study discontinuation are reported in the Participant Flow section. All deaths regardless of causality or whether they were reported as a reason for study discontinuation are reported in the All-Cause Mortality section.) | 0 | 0 | 23
Not Completed | 3 | 3 | 33
Not completed — Physician Decision | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 6
Not completed — Participant excluded from efficacy population | 0 | 0 | 1
Not completed — Death | 0 | 0 | 2
Not completed — Progressive Disease | 2 | 2 | 2
Not completed — Disease progression needing additional medication | 0 | 0 | 17
Not completed — Sponsor decision | 0 | 0 | 2
Not completed — Other Medical Reasons | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 dose of MEN1611.
Groups:
- Dose Expansion Cohort: Participants received high dose of MEN1611 (RP2D) twice daily administered in combination with trastuzumab once every 3 weeks ± fulvestrant once every 4 weeks.
- Total: Total of all reporting groups
Arm/Group | Dose Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Expansion Cohort | Total
Number analyzed (Participants) | 3 | 3 | 56 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 43 | 46
  >=65 years | 2 | 1 | 13 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (7.937) | 59.33 (14.468) | 53.36 (11.112) | 56.02 (55.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 56 | 62
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 3 | 3 | 50 | 56
  Unknown | 0 | 0 | 5 | 5

OUTCOME MEASURES:

1. Primary Outcome: MTD of MEN1611 in Combination With Trastuzumab ± Fulvestrant
Description: MTD was defined as the highest dose level at which no more than 1 participant experienced a DLT during the 28-day DLT assessment window.
Time Frame: Up to 28 Days
Population: DLT population included all participants from Dose Escalation Cohorts 1, 2 and 3 participants from the Dose Expansion Cohort.
  DLT population consisted of all participants who received at least 80% of MEN1611 and 100% of trastuzumab and/or fulvestrant during 28 days after the first MEN1611 drug administration with a Safety Follow-up of 28 days after the first administration of the study treatment.
Measure: Number; unit: milligrams (mg)
Groups:
- Dose Escalation Cohorts 1 and 2, and Dose Expansion Cohort: Participants received low, medium, or high dose of MEN1611 respectively, twice daily administered in combination with trastuzumab once every 3 weeks ± fulvestrant once every 4 weeks.
Arm/Group | Dose Escalation Cohorts 1 and 2, and Dose Expansion Cohort
Number analyzed (Participants) | 9
milligrams (mg) | 48

2. Primary Outcome: Number of Participants With DLTs of MEN1611 in Combination With Trastuzumab ± Fulvestrant
Description: DLT was defined as the occurrence of any of the protocol defined adverse drug reactions (ADRs) related to the combination regimens or to MEN1611 alone and unrelated to the participants' underlying disease or concomitant medication occurring during 28 days after the first MEN1611 administration.
Time Frame: Up to 28 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Dose Escalation Cohort 3: Participants received high dose of MEN1611 (RP2D) twice daily administered in combination with trastuzumab once every 3 weeks ± fulvestrant once every 4 weeks.
Arm/Group | Dose Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3
Number analyzed (Participants) | 3 | 3 | 3
Participants | 0 | 0 | 0

3. Primary Outcome: RP2D of MEN1611 in Combination With Trastuzumab ± Fulvestrant
Description: RP2D was defined as the highest dose level in milligrams (mg) at which no more than 1 participant experienced a DLT during the DLT assessment window (28days), or the maximum dose judged to be tolerable.
Time Frame: Up to 28 days
Population: as for outcome 1
Measure: Number; unit: mg
Arm/Group | Dose Escalation Cohorts 1 and 2, and Dose Expansion Cohort
Number analyzed (Participants) | 9
mg | 48

4. Secondary Outcome: Best Overall Response (BOR) of MEN1611 in Combination With Trastuzumab ± Fulvestrant
Description: BOR was defined as percentage of participants who had a best overall response to therapy of complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD) and was defined according to Response Evaluation Criteria in Solid Tumors version 1.1 assessment locally performed using computed tomography scans or magnetic resonance imaging of the chest and abdomen (including pelvis and adrenal glands).
Time Frame: Up to 3 years
Population: Efficacy Population included all eligible participants who received at least 8 weeks of any treatment and had at least 1 disease assessment. Here, 'Overall Number of Participants Analyzed' = participants who were evaluable for this Outcome Measure.
Measure: Number; unit: percentage of participants
Arm/Group | Dose Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Expansion Cohort
Number analyzed (Participants) | 3 | 3 | 42
percentage of participants
  Complete Response (CR) | 0 | 0 | 4.8
  Partial Response (PR) | 0 | 66.7 | 35.7
  Stable Disease (SD) | 33.3 | 33.3 | 47.6
  Non-CR/Non-PD | 0 | 0 | 0
  Progressive Disease (PD) | 66.7 | 0 | 9.5
  Not Evaluable (NE) | 0 | 0 | 2.4

5. Secondary Outcome: Objective Response Rate (ORR) of MEN1611 in Combination With Trastuzumab ± Fulvestrant
Description: ORR was calculated as the sum of the Best Overall Response (BOR) of complete response (CR) and partial response (PR) rates. ORR was defined according to Response Evaluation Criteria in Solid Tumors version 1.1assessment performed using computed tomography scans or magnetic resonance imaging of the chest and abdomen (including pelvis and adrenal glands).
Time Frame: Up to 3 years
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Expansion Cohort
Number analyzed (Participants) | 3 | 3 | 42
percentage of participants | 0 [0 to 70.8] | 66.7 [9.4 to 99.2] | 40.5 [25.6 to 56.7]

6. Secondary Outcome: Disease Control Rate (DCR) of MEN1611 in Combination With Trastuzumab ± Fulvestrant
Description: DCR was defined as percentage of participants whose disease shrank or remained stable over a certain time period and was calculated as the sum of the best overall response (BOR) rates of CR, PR and Stable Disease (SD) rates.
Time Frame: Up to 3 years
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Expansion Cohort
Number analyzed (Participants) | 3 | 3 | 42
percentage of participants | 33.3 [0.8 to 90.6] | 100 [29.2 to 100] | 88.1 [74.4 to 96]

7. Secondary Outcome: Duration of Response (DOR) of MEN1611 in Combination With Trastuzumab ± Fulvestrant
Description: DOR was defined as time from first occurrence of a BOR of PR, CR or SD as locally assessed, until the disease has been shown to progress following treatment. Participants with a previous response who did not show a relapse or die without recording a relapse were censored at their last available relapse-free tumour assessment date. Participants with only one tumour assessment after baseline showing progressive disease (PD) were not included in the calculation.
Time Frame: Up to 3 years
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Dose Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Expansion Cohort
Number analyzed (Participants) | 3 | 3 | 42
days | 224 [0 to NA] — Upper confidence interval (CI) not calculable due to an insufficient number of participants with events. | NA [29 to NA] — Median and Upper CI not calculable due to an insufficient number of participants with events. | 114 [65 to 244]

8. Secondary Outcome: Progression-free Survival (PFS) of MEN1611 in Combination With Trastuzumab ± Fulvestrant
Description: PFS was defined as the number of days between the first study treatment administration to the date of first documented disease progression as per local assessment, relapse or death from any cause. Responding participants and participants who were lost to follow-up were censored at their last tumour assessment date.
Time Frame: Up to 3 years
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Dose Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Expansion Cohort
Number analyzed (Participants) | 3 | 3 | 42
days | 62 [53 to NA] — Upper CI not calculable due to an insufficient number of participants with events. | 203 [106 to NA] — Upper CI not calculable due to an insufficient number of participants with events. | 167 [116 to 217]

9. Secondary Outcome: Overall Survival (OS) of MEN1611 in Combination With Trastuzumab ± Fulvestrant
Description: OS was defined as the number of days between the first study treatment administration and death from any cause. Participants still alive who had withdrawn from the study were censored using the latest among end of study and follow-up dates. Drop-out participants were considered censored and the last available date in which the participant was known to be alive were used for calculation.
Time Frame: Up to 3 years
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Dose Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Expansion Cohort
Number analyzed (Participants) | 3 | 3 | 28
days | 120 [112 to NA] — Upper CI not calculable due to an insufficient number of participants with events. | 203 [143 to NA] — Upper CI not calculable due to an insufficient number of participants with events. | 989 [513 to NA] — Upper CI not calculable due to an insufficient number of participants with events.

ADVERSE EVENTS:
Time Frame: Up to approximately 3 years
Description: Safety Population included all participants who received at least 1 dose of MEN1611.
  All deaths regardless of causality or whether they were reported as a reason for study discontinuation are reported in the All-Cause Mortality section. Only deaths notified as leading to study discontinuation are reported in the Participant Flow section.
  Deaths that occurred during the follow-up after completion of the treatment period were collected for all cohorts.
Arm/Group | Dose Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Expansion Cohort
All-Cause Mortality (participants affected / at risk) | 3/3 | 3/3 | 28/56
Serious Adverse Events (participants affected / at risk) | 2/3 | 3/3 | 21/56
Other Adverse Events (participants affected / at risk) | 2/3 | 3/3 | 56/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation Cohort 1 (N=3) | Dose Escalation Cohort 2 (N=3) | Dose Expansion Cohort (N=56)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 3
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 0 | 1 | 0
General physical health deterioration (General disorders) | 0 | 0 | 1
Generalised oedema (General disorders) | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 2
Pneumonia (Infections and infestations) | 0 | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 0 | 1
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lipase increased (Investigations) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Brachial plexopathy (Nervous system disorders) | 0 | 0 | 1
Facial nerve disorder (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1
Paraparesis (Nervous system disorders) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation Cohort 1 (N=3) | Dose Escalation Cohort 2 (N=3) | Dose Expansion Cohort (N=56)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 18
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 5
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 5
Blepharitis (Cardiac disorders) | 0 | 0 | 3
Dry eye (Cardiac disorders) | 0 | 0 | 4
Xerophthalmia (Cardiac disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 6
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 5
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 6
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 36
Discoloured vomit (Gastrointestinal disorders) | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 6
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 5
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 2
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 4
Nausea (Gastrointestinal disorders) | 2 | 0 | 26
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 11
Vomiting (Gastrointestinal disorders) | 0 | 0 | 14
Asthenia (General disorders) | 1 | 3 | 15
Fatigue (General disorders) | 0 | 0 | 6
Influenza like illness (General disorders) | 0 | 0 | 3
Mucosal inflammation (General disorders) | 0 | 1 | 9
Oedema peripheral (General disorders) | 1 | 1 | 10
Pyrexia (General disorders) | 0 | 0 | 15
Temperature regulation disorder (General disorders) | 0 | 1 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 3
COVID-19 (Infections and infestations) | 0 | 0 | 4
Conjunctivitis (Infections and infestations) | 0 | 1 | 2
Paronychia (Infections and infestations) | 0 | 1 | 3
Pneumonia (Infections and infestations) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 7
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 2
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 11
Amylase increased (Investigations) | 0 | 1 | 7
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 12
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 5
Blood bilirubin increased (Investigations) | 0 | 1 | 5
Blood creatinine increased (Investigations) | 0 | 0 | 3
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 4
Blood phosphorus decreased (Investigations) | 0 | 1 | 1
Ejection fraction decreased (Investigations) | 0 | 0 | 5
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 6
Glycosylated haemoglobin increased (Investigations) | 0 | 0 | 3
Lipase increased (Investigations) | 0 | 1 | 8
Lymphocyte count decreased (Investigations) | 0 | 0 | 4
Weight decreased (Investigations) | 0 | 0 | 5
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 14
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 21
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 5
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 7
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 3
Polydipsia (Metabolism and nutrition disorders) | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 6
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 2
Dysarthria (Nervous system disorders) | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 9
Headache (Nervous system disorders) | 0 | 0 | 11
Sciatica (Nervous system disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 3
Dysuria (Renal and urinary disorders) | 0 | 1 | 1
Polyuria (Renal and urinary disorders) | 0 | 1 | 2
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 1 | 0
Vulvovaginal inflammation (Reproductive system and breast disorders) | 0 | 1 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 6
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 15
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Haematoma (Vascular disorders) | 1 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 5
Lymphoedema (Vascular disorders) | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the study cannot be submitted for presentation, abstract, poster exhibition, or publication by the investigator until Menarini Ricerche S.p.A. has reviewed/commented and agreed to any publication.

DOCUMENTS (2):
  • Study Protocol (2022-03-03): https://cdn.clinicaltrials.gov/large-docs/35/NCT03767335/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-11): https://cdn.clinicaltrials.gov/large-docs/35/NCT03767335/SAP_001.pdf